CLINICAL TRIAL: NCT07342283
Title: QL1706 Plus Chemotherapy as Neoadjuvant Therapy in Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K223-02
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): QL1706 plus carboplatin and albumin-bound paclitaxel (21-day cycles for 4 cycles) followed by QL1706 plus doxorubicin/epirubicin and cyclophosphamide (21-day cycles for 4 cycles)
  Interventions: Drug: Immunotherapy combined with chemotherapy

INTERVENTIONS:
Drug: Immunotherapy combined with chemotherapy — Albumin-bound paclitaxel: 125 mg/m², day 1 and day 8, 21-day cycle; Carboplatin: AUC = 5, day 1 or AUC = 2-3, day 1 and day 8, 21-day cycle; QL1706: 5 mg/kg, day 1, 21-day cycle; Epirubicin: 90-100 mg/m², day 1, 21-day cycle; or Doxorubicin: 50 mg/m², day 1, 21-day cycle; Cyclophosphamide: 600 mg/m², day 1, 21-day cycle.

SUMMARY:
This is a single-center, single-arm, prospective study enrolling 30 patients with stage II-III triple-negative breast cancer. The neoadjuvant regimen consists of QL1706 combined with carboplatin plus albumin-bound paclitaxel (21-day cycles for 4 cycles) followed by QL1706 combined with doxorubicin/epirubicin plus cyclophosphamide (21-day cycles for 4 cycles). The treatment observation period is 1 year, and the primary endpoint is the pathological complete response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed newly diagnosed ER-/HER2- breast cancer. ER and PR with Allred score <3 or <1% positively stained cells in tumor infiltrating components. HER2 negativity defined as 0 or 1+ by FISH or IHC staining per NCCN guidelines;
2. Clinical stage II or III breast cancer eligible for neoadjuvant chemotherapy (per AJCC 8th edition: at least T2 any N M0, or any T if N+), with treatment goal of complete surgical resection following neoadjuvant therapy;
3. Tumor size ≥2 cm by clinical or imaging assessment per WHO criteria. Patients with histologically confirmed or clinically palpable lymph nodes are eligible regardless of tumor size;
4. Treatment-naïve subjects;
5. Age ≥18 years, both genders eligible;
6. ECOG performance status 0-1;
7. Adequate bone marrow, cardiac, and organ function;
8. Women of childbearing potential must have a negative pregnancy test (serum or urine HCG) within 30 days prior to study enrollment and must practice effective contraception during the study;
9. Ability to comprehend and provide written informed consent.

Exclusion Criteria:

1. History of invasive malignancies within 5 years prior to signing the informed consent form, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or carcinoma in situ of the cervix;
2. Subjects who have received chemotherapy, immunotherapy, targeted therapy, or radiotherapy within the past 12 months;
3. Stage IV metastatic breast cancer;
4. Administration of a vaccine within 30 days before the first dose of the study treatment;
5. Subjects with severe systemic diseases;
6. Subjects with active infections (including but not limited to HIV, hepatitis B or C, tuberculosis);
7. Severe cardiovascular diseases, such as: history of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass grafting within the past 6 months; or congestive heart failure (CHF) of New York Heart Association (NYHA) class II-IV, or history of CHF NYHA class III or IV;
8. Lactating women should discontinue breastfeeding during the study;
9. Subjects with known allergies to the study drug or any of its excipients;
10. Any other condition deemed inappropriate for participation in the study by the investigator.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rates | Up to approximately 9 months
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Objective response rate（ORR） | Up to approximately 27-30 weeks
  Percentage of Participants With an Objective Response of CR or PR According to RECIST v1.1
3y-EFS | Up to approximately 3 years
  Percentage of patients who, from the initiation of treatment, remain free of any of the following events within three years: disease progression to unresectable status, local or distant recurrence, development of a second primary malignancy (breast cancer or other cancers), or death from any cause.
Overall survival (OS) | Up to approximately 8 years
  OS is defined as the time from the initiation of treatment to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.
Adverse events | up to 18 months
  AEs will be assessed according to NCI CTCAE v5.0, by grade

IPD SHARING:
Plan to Share IPD: No